CLINICAL TRIAL: NCT07380139
Title: Dexamethasone Versus Dexmedetomidine as Adjuvant to Bupivacaine in Sphenopalatine Ganglion Block as Post-operative Analgesia in Rhinoplasty Surgeries
Brief Title: Dexamethasone vs Dexmedetomidine in Sphenopalatine Ganglion Block for Rhinoplasty Pain
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MD255/2025
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group B (Active Comparator): Group B (control group): will receive bupivacaine 0.25% (3ml) + normal saline, total volume (5 ml).
  Interventions: Drug: Bubpivacaine
- Group BDX (Active Comparator): Group BDX: will receive bupivacaine 0.25% (3ml) + dexmedetomidine (1 mic/kg), total volume 5ml by adding normal saline.
  Interventions: Drug: Dexamedomedine
- Group BD (Active Comparator): Group BD: will receive bupivacaine 0.25% (3ml) + dexamethasone (4mg), total volume 5ml by adding normal saline
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamedomedine — will receive bupivacaine 0.25% (3ml) + dexmedetomidine (1 mic/kg), total volume 5ml by adding normal saline.
  Arms: Group BDX
Drug: Dexamethasone — will receive bupivacaine 0.25% (3ml) + dexamethasone (4mg), total volume 5ml by adding normal saline
  Arms: Group BD
Drug: Bubpivacaine — will receive bupivacaine 0.25% (3ml) + normal saline, total volume (5 ml).
  Arms: Group B

SUMMARY:
This study will test the effect of adding dexamethasone versus dexmedetomidine as adjuvants to bupivacaine in sphenopalatine ganglion block used for pain after rhinoplasty

DETAILED DESCRIPTION:
Preoperative settings:

Preoperative evaluation of full medical history will be taken, examination will be done, and routine preoperative investigations will be done to all patients including complete blood picture and coagulation profile.

The patient will be fasting for at least 8 hours preoperatively

Intraoperative settings:

General anesthesia technique:

Upon arrival to OR, Standard monitoring will be applied: ECG, non-invasive blood pressure and pulse oximeter, Intravenous access (20G) will be inserted, and all patients will receive midazolam 0.05mg/kg IV for anxiety, ranitidine 50 mg IV and ondansetron 0.15mg/kg IV 15 min before induction.

Induction of anesthesia in all groups will be done by intravenous propofol 2-2.5 mg/kg IV, fentanyl 1 µg/kg IV and atracurium 0.5 mg/kg IV, then endotracheal tube of suitable size will be applied and capnogram will be connected. Maintenance will be achieved by isoflurane inhalation started with 1.2 % and top-up doses of atracurium (0.01 mg/kg IV). Volume controlled positive pressure ventilation was adjusted at tidal volume and respiratory rate to keep ETCO2 at 35-40 mmHg with continuous monitoring. During surgery, the patients received intravenous infusion of ringer solution according to fluid requirement regimen. Fluid administration will be guided by hemodynamics monitoring and clinical parameters

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Sex: of either sex.
3. American Society of Anaesthesiologists (ASA) Physical Status Class I and II.
4. BMI < 35
5. Scheduled for rhinoplasty surgeries under general anaesthesia.

Exclusion Criteria:

1. Declining to give written informed consent.
2. History of allergy to the medications used in the study.
3. Contraindications to regional anesthesia (including patient refusal, coagulopathy and local infection).
4. Psychiatric disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The time to the first request of analgesia | 9 months
  The time interval between the onset of the local infiltration done at the end of the operation and the first request to postoperative analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided